CLINICAL TRIAL: NCT06137105
Title: A Study of Treatment With Thrombopoietin Agonists in Patients With Idiopathic Thrombocytopenic Purpura
Brief Title: Thrombopoietin Agonists in Patients With Idiopathic Thrombocytopenic Purpura
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Responsible Party: Principal Investigator, Naira Ibrahem Ahmed Saad, A Study of Treatment with thrombopoietin agonists in patients with Idiopathic thrombocytopenic purpura, Assiut University
Other Study IDs: TPO in ITP
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group I : Romiplostim and Eltrombopag
  Interventions: Drug: eltrombopag and romiplastim
- Group 2: Group II : recived corticosteroid.
  Interventions: Drug: eltrombopag and romiplastim

INTERVENTIONS:
Drug: eltrombopag and romiplastim — Group I: eltrombopag and romiplastim
  Group II : recived corticosteroid.
  Other Names: Corticosteroids

SUMMARY:
1. Assesement of response to Thrombopoietin receptor agonists (TPO-RAs) as treatment in Idiopathic thrombocytopenia purpura patients in Assiut University hospital.
2. Explore side effects of Thrombopoietin receptor agonists in Idiopathic thrombocytopenia purpura .
3. To study effect of thrombopoietin receptor agonists and Quality life in Idiopathic thrombocytopenia purpura patients.

DETAILED DESCRIPTION:
Idiopathic thrombocytopenic purpura (ITP) is an autoimmune disorder characterized by reduced platelet counts (<100 × 109/L) and increased bleeding risk in the absence of other causes associated with thrombocytopenia().. It affects 2-4 per 100,000 individuals annually with an overall prevalence of about 10/100,000 individuals().

Manifestations of idiopathic thrombocytopenic purpura( ITP) can be localised haemorrhaging in skin or mucous membranes that are usually of little to no clinical consequence (petechiae, purpura, ecchymoses, epistaxis); more rarely, ITP can be associated with severe bleeding events such as intracranial haemorrhage (ICH). However, most ITP patients are asymptomatic in the presence of platelet counts greater than 50x109/L2.()

Idiopathic thrombocytopenia purpura is diagnosed in absence of secondary causes of immune mediated thrombocytopenia including autoimmune diseases (systemic lupus erthematosus , antiphospholipid antibody syndrome) lymphoproliferative disorders (chronic lymphocytic leukemia ) viral infection (hepatitis c virus , human immunodeficiency virus

The goal of treatment in patients with of idiopathic thrombocytopenic purpura is to maintain the platelet count at a level that reduces the risk of bleeding with minimal treatment-related toxic effects. Observation alone is recommended when no or mild bleeding is present and the platelet count is more than 30,000 per cubic millimeter in adults.23 Treatment in patients with a lower platelet count is indicated only if bleeding occurs or if the platelet count is very low. (For example, most experts would treat a non bleeding patient who had a platelet count of <10,000 per cubic millimeter().

Historically , the treatment of idiopathic thrombocytopenia purpura has been directed at inhibiting the production of anti platelet autoantibodies or opsonization of antibody coated platelets. However, impaired platelet production is increasingly recongnized as a contributor to thrombocytopenia in patients with idiopathic thrombocytopenia purpura.

New treatment guidelines have supported a shift from corticosteroids and splenectomy to newer medical treatments that mitigate the thrombocytopenia and avoid splenectomy. The thrombopoietin receptor agonists (TPO-RA), romiplostim, eltrombopag, and avatrombopag, have markedly altered the treatment of ITP()

Thrombopoietin (TPO) is the main cytokine that stimulates thrombopoiesis, and although platelet counts are low in ITP patients, no compensatory increase in TPO production occurs in these patients().

Thrombopoietin receptor agonists (TPO-RAs) are TPO mimetics that can bind to and activate TPO receptors, leading to megakaryocyte maturation, proliferation and differentiation and resulting in increased platelet production. Two major TPO-RAs, romiplostim and eltrombopag, have been investigated in several randomized controlled trials (RCTs) involving adult and pediatric ITP patients the results of which are encouraging. Currently, romiplostim and eltrombopag are recommended as second-line therapeutic options for adult ITP patients().

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with Idiopathic thrombocytopenic purpura (ITP)

  1. patients above age of 18 years.

Exclusion Criteria:

* patients below age of 18 years .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presented with Idiopathic thrombocytopenic purpura ( ITP) at clinical Hematology units, Internal Medicine Department at Assiut University .
  Patients above age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of response to treatment will be clinical and laboratory assessment | Baseline
  Platelet count should be measured weekly until a stable platelet count that is associated with an absence of bleeding symptoms is achieved for 4 weeks without adjustment and then measured monthly thereafter.